CLINICAL TRIAL: NCT05239637
Title: A Randomized Controlled Pilot Trial of When Heparin Stopped for Anticoagulation During Extracorporeal Membrane Oxygenation Decannulation
Brief Title: When Heparin Stopped for Anticoagulation During ECMO Decannulation
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Second Affiliated Hospital of Zhengzhou University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: LHGJ20210421
Record Dates: First submitted 2021-12-21; First posted 2022-02-15 (Actual); Last update posted 2022-03-15 (Actual); Status verified 2022-02

CONDITIONS: Extracorporeal Membrane Oxygenation
Keywords: Extracorporeal Membrane Oxygenation; Heparin; Anticoagulants; Decannulation; Randomized Controlled

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Previous (Experimental): Heparin stopped before ECMO decannulation
  Interventions: Other: Heparin stopped before ECMO decannulation
- Afterwards (Experimental): Heparin reduced after ECMO decannulation
  Interventions: Other: Heparin reduced after ECMO decannulation

INTERVENTIONS:
Other: Heparin stopped before ECMO decannulation — Heparin has been stopped for 1 hour before ECMO decannulation;The cannulas can be removed immediately with clots larger than 5 mm or enlarging clots in the circuit.
  Arms: Previous
Other: Heparin reduced after ECMO decannulation — Heparin gradually reduced within 24 hours after ECMO decannulation, If excess bleeding occured,decrease the heparin infusion rapidly or turn the heparin off immediately. Protamine can be given to reversing heparin if necessary.
  Arms: Afterwards

SUMMARY:
Heparin (regular or unfractionated heparin, not low molecular weight heparin) is given as a bolus (50-100 units per kilogram) at the time of extracorporeal membrane oxygenation(ECMO) cannulation, and by continuous infusion during ECMO. Heparin infusion is regulated to keep the whole blood activated clotting time (ACT) or activated partial thromboplastin time (APTT) at a designated level (usually 1.5 times normal for the ACT or APTT measurement system). An elevated ACT or APTT is associated with high risks of early and late complications,such as bleeding,hematoma,pseudoaneurysm,and arterial-venous fistula. Extracorporeal life support organization(ELSO) make recommendation that the cannulas can be removed ideally after the heparin has been stopped for 30 to 60 minutes.However,the Chinese Thoracis Society recommends that heparin should not be discontinued immediately before ECMO decannulation, but gradually reduced within 24 hours, and then low molecular weight heparin is continued to be given for anticoagulation. Therefore,options of which time heparin stopped remain controversial.The investigators conduct this pilot study to investigate the opportunity of heparin stopped for anticoagulation before ECMO decannulation.

DETAILED DESCRIPTION:
Forty adult patients with cardiac or respiratory failure supported by ECMO are enrolled in the study. Patients are randomly allocated to be treated with either a) heparin has been stopped for 1 hour before ECMO decannulation(regimen A), b) heparin gradually reduced within 24 hours after ECMO decannulation(regimen B).The investigators hypothesize that patients treated with regimen A as compared with patients treated with regimen B would decrease the incidence of complications during the ECMO decannulation period(from 1 hour before ECMO decannulation to 72 hours post decannulation).

ELIGIBILITY:
Inclusion Criteria:

* ECMO therapy was instituted to support circulatory and/or respiratory failure;
* Heparin continuous infusion for anticoagulation during ECMO;
* Native cardiac and pulmonary function improve,and the trial off is successful.
* Ensure each patient provides signed and dated informed consent.

Exclusion Criteria:

* 1.History of thrombotic diseases or coagulation disorder；
* Thrombosis or bleeding events occurred prior to allocation；
* Heparin stopped prior to allocation；
* Other anticoagulants, antiplatelets, hemostatics and other drugs affected coagulation function have been used；
* The trial off has failed;
* Pregnant and lactating patients;
* Patients participated in the other studies;
* Patients couldn't accept comprehensive treatment;
* Patients couldn't acquire informed consent;

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2022-02-15 (Actual); Primary Completion 2023-10 (Estimated); Study Completion 2023-10 (Estimated)

PRIMARY OUTCOMES:
Incidence of bleeding and clotting complications | 72 hours after decannulation

SECONDARY OUTCOMES:
ICU mortality | 1 day after ICU discharge
28-days mortality | 28 days after decannulation
Prothrombin time | 1 day and 3 days after decannulation
  Measured at the laboratory
Activated partial thromboplastin time | 1 day and 3 days after decannulation
  Measured at the laboratory
International normalised ratio | 1 day and 3 days after decannulation
  Measured at the laboratory
Fibrinogen | 1 day and 3 days after decannulation
  Measured at the laboratory
D-dimer | 1 day and 3 days after decannulation
  Measured at the laboratory
R time | 1 day and 3 days after decannulation
  Time to initial fibrin formation in minutes
K time | 1 day and 3 days after decannulation
  Minutes to 20 mm clot strength
α angle | 1 day and 3 days after decannulation
  Rate of clot strengthening
Maximum amplitude（MA） | 1 day and 3 days after decannulation
  MA represents the ultimate strength of the fibrin clot in mm
LY30 | 1 day and 3 days after decannulation
  Degree of clot lysis at 30 minutes
Volume of packed red cells transfusion | 3 days after decannulation

CONTACTS AND LOCATIONS:
Overall Officials: Li yahui, Master, Principal Investigator — Second Affiliated Hospital of Zhengzhou University
Locations (1):
- General ICU of the second affiliated hospital of zhengzhou university, Zhengzhou, Henan, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Tonna JE, Abrams D, Brodie D, Greenwood JC, Rubio Mateo-Sidron JA, Usman A, Fan E. Management of Adult Patients Supported with Venovenous Extracorporeal Membrane Oxygenation (VV ECMO): Guideline from the Extracorporeal Life Support Organization (ELSO). ASAIO J. 2021 Jun 1;67(6):601-610. doi: 10.1097/MAT.0000000000001432. PMID 33965970
- See also: The chinese thoracis society recommended that heparin should not be discontinued immediately before ECMO decannulation — http://rs.yiigle.com/CN112147201909/1161183.htm